CLINICAL TRIAL: NCT03201016
Title: Prevalence of Osteoporosis and Fractures in Patients With Hepatic Cirrhosis and Investigation of the Associated Factors
Acronym: POC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Jordi Sanchez-Delgado, Jordi Sánchez Delgado M.D; PhD. Staff of the Hepatology Unit. Digestive Diseases Department. Principal Investigator, Corporacion Parc Tauli
Other Study IDs: 2015540
Record Dates: First submitted 2017-05-09; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Osteoporosis
Keywords: cirrhosis
MeSH Terms: conditions — Osteoporosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bone densitometry — Procollagen Type I Propeptides, alkaline phosphatase, Crosslinked Telopeptides of Type I Collagen
  Other Names: Trabecular Bone Score

SUMMARY:
Osteoporosis is a common complication in chronic liver disease, especially in the late stages of the disease. Good nutrition and calcium and vitamin D supplementation are recommended for the prevention and treatment of osteoporosis. There are no specific guidelines for its pharmacological treatment, but bisphosphonates have been shown to be effective in increasing bone mass in patients with chronic cholestasis, with a good safety profile.

There are few studies evaluating the prevalence of osteoporosis in patients with cirrhosis (except for primary biliary cholangitis (PBC)). There are no clear recommendations for osteoporosis screening in cirrhotic patients. A diagnosis and early therapeutic intervention before the onset of the complications derived would significantly improve the quality of life and decrease the morbidity and mortality associated with osteoporosis and fractures

Objective:

-To assess the prevalence of osteoporosis and fragility fractures in patients with liver cirrhosis in our country and the risk factors associated

Method:

Patients diagnosed with hepatic cirrhosis, other than PBC, will be included in any Child stage during a hospital admission. Epidemiological, demographic, clinical, analytical and imaging data (dorso-lumbar spine radiography, bone densitometry and Trabecular Bone Score) will be evaluated. A descriptive statistic of the main variables will be carried out as well as a multivariate analysis to evaluate the predictive factors of osteoporosis and / or fragility fractures

DETAILED DESCRIPTION:
Osteoporosis is a common complication in chronic liver disease, especially in the late stages of the disease. The main mechanism involved in the development of osteoporosis in patients with cirrhosis is the deficit of bone formation due to the harmful effect of substances such as bilirubin and bile acids or the toxic effect of alcohol or iron on osteoblasts .

Good nutrition and calcium and vitamin D supplementation are recommended for the prevention and treatment of osteoporosis. There are no specific guidelines for its pharmacological treatment, but bisphosphonates have been shown to be effective in increasing bone mass in patients with chronic cholestasis, with a good safety profile.

Hospital admissions in relation to osteoporotic fractures in cirrhotic patients are frequent with a high morbidity and mortality rate. There are few studies evaluating the prevalence of osteoporosis in patients with cirrhosis with a different etiology from PBC and the existing series are published years ago with few patient numbers. There are no clear recommendations for osteoporosis screening in cirrhotic patients. A diagnosis and early therapeutic intervention before the onset of the complications derived would significantly improve the quality of life and decrease the morbidity and mortality associated with osteoporosis and fractures

Objective:

* To assess the prevalence of osteoporosis and fragility fractures in patients with liver cirrhosis in our country.
* To assess the risk factors associated with osteoporosis and fractures in these patients.

Method:

Patients diagnosed with hepatic cirrhosis, other than PBC, will be included in any Child stage during a hospital admission. Epidemiological, demographic, clinical, analytical and imaging data (dorso-lumbar spine radiography, bone densitometry and Trabecular Bone Score) will be evaluated. Additional visits to those already carried out in normal practice will not be necessary. A descriptive statistic of the main variables will be carried out as well as a multivariate analysis to evaluate the predictive factors of osteoporosis and / or fragility fractures

ELIGIBILITY:
Inclusion Criteria:

* Give informed consent to participate in the study
* Hepatic cirrhosis diagnosed by histological criteria or clinical, analytical and ultrasound criteria
* Age over 18 years

Exclusion Criteria:

* Ascitic decompensation (estimated ascitic fluid> 4 liters) at the time of bone densitometry
* Patients bedridden or with very bad mobility, that makes the displacement complicated
* Terminal illness with estimated life expectancy less than one year due to hepatic impairment or tumor disease

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with hepatic cirrhosis due to hepatitis C virus or alcohol, decompensated or not decompensated and who follow controls in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Assess the prevalence of osteoporosis and fractures in patients with hepatic cirrhosis | It is a cross-sectional prevalence study. Patients will be recruited for two years.
  To confirm the presence of osteoporosis and fractures in patients with cirrhosis, the investigators wil perform:
  - Bone Densitometry measured in standard deviations

SECONDARY OUTCOMES:
Assess the associated factors risk of osteoporosis and fractures | It is a cross-sectional prevalence study. Patients will be recruited for two years.
  Factors that will be studied:
  • Data regarding cirrhosis (etiology; alcohol/hepatitis C virus, both of them)

OTHER OUTCOMES:
Assess the prevalence of osteoporosis and fractures using trabecular bone score | It is a cross- sectional prevalence study. Patients will be recruited for two years.
  The TBS (Trabecular Bone Score) is derived from the evaluation of the experimental variogram, obtained from the grayscale of the bone densitometry. This score may be more sensitive to detect osteoporosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Sánchez-Delgado, M.D. PhD, Principal Investigator — Unitat de Malalties Digestives, Parc Taulí Hospital Universitari, Institut d'Investigació i Innovació Parc Taulí I3PT
Locations (1):
- Corporació Sanitària i Universitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No